CLINICAL TRIAL: NCT02367898
Title: Enhancing Cognitive Abilities With Comprehensive Training: A Large, Online, Randomized, Active-Controlled Trial
Brief Title: Enhancing Cognitive Abilities With Comprehensive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumos Labs, Inc. (Industry)
Collaborators: Wheaton College (Other); Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: LLI-001
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Cognitive Abilities
Keywords: Cognitive Training; Lumosity; Crossword Puzzles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Training (Experimental): Lumosity cognitive training program.
  Interventions: Other: Lumosity Cognitive Training
- Crossword Puzzles (Active Comparator): Timed online crossword puzzles
  Interventions: Other: Crossword Puzzles

INTERVENTIONS:
Other: Lumosity Cognitive Training — adaptive online cognitive training
  Arms: Cognitive Training
Other: Crossword Puzzles — timed online crossword puzzles
  Arms: Crossword Puzzles

SUMMARY:
The purpose of this study is to measure the efficacy of an online cognitive training program against an active control condition in a large, randomized trial.

DETAILED DESCRIPTION:
The present study aims to evaluate a targeted, progressively challenging, online cognitive training program comprised of 49 distinct exercises targeting a variety of cognitive capacities. The cognitive training program will be compared to a plausibly beneficial active control condition in which participants completed online crossword puzzles.

The investigators hypothesize that the cognitive training will show greater transfer to a range of underlying cognitive abilities than the active control, as measured by a broad battery of neuropsychological assessments and participant-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Engaged with the Lumosity program at least 3 days in the first week after sign-up
* Access to an internet enabled computer to complete training

Exclusion Criteria:

* Paying subscriber

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11470 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Aggregate Cognitive Performance | Baseline to 10 weeks
  Aggregate cognitive performance, as measured by Grand Index, on seven neuropsychological assessments (Forward Memory Span, Reverse Memory Span, Grammatical Reasoning, Progressive Matrices, Go/No-Go, Arithmetic Reasoning, Two-Target Search)

SECONDARY OUTCOMES:
Participant-Reported Outcomes | Baseline to 10 weeks
  9 questions related to everyday cognition and emotional status.
Individual Neuropsychological Assessments composite | Baseline to 10 weeks
  Separate analyses of changes on each of the seven neuropsychological assessments in the battery (Forward Memory Span, Reverse Memory Span, Grammatical Reasoning, Progressive Matrices, Go/No-Go, Arithmetic Reasoning, Two-Target Search).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sternberg, PhD, Principal Investigator — Lumos Labs, Inc.
Locations (1):
- Lumos Labs, Inc., San Francisco, California, United States

REFERENCES:
- [Derived] Hardy JL, Nelson RA, Thomason ME, Sternberg DA, Katovich K, Farzin F, Scanlon M. Enhancing Cognitive Abilities with Comprehensive Training: A Large, Online, Randomized, Active-Controlled Trial. PLoS One. 2015 Sep 2;10(9):e0134467. doi: 10.1371/journal.pone.0134467. eCollection 2015. PMID 26333022
- See also: Click here for more information about Lumosity's Human Cognition Project. — http://www.Lumosity.com/hcp